CLINICAL TRIAL: NCT01108627
Title: Effect of Gly16Arg Polymorphism in ADRB2 Gene on Asthma Control in Children Receiving Long Acting Beta Agonists
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Drug supply sponsor sent outdated drug
Sponsor: Nemours Children's Clinic (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 3203534014
Record Dates: First submitted 2010-04-19; First posted 2010-04-22 (Estimated); Last update posted 2023-05-26 (Actual); Status verified 2023-05

CONDITIONS: Safety of Long Acting Beta Agnoists
MeSH Terms: interventions — Formoterol Fumarate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- corticosteroid + long acting beta agonist; steroids (Active Comparator)
  Interventions: Drug: open-labeled inhaled corticosteroids (ICS); FORADIL® AEROLIZER®; Drug: foradil
- placebo + corticosteroid + long acting beta agonist; steroids (Placebo Comparator)
  Interventions: Drug: foradil placebo

INTERVENTIONS:
Drug: open-labeled inhaled corticosteroids (ICS); FORADIL® AEROLIZER® — • Drugs. The study drugs are open-labeled inhaled corticosteroids (ICS); FORADIL® AEROLIZER® and FORADIL placebo. FORADIL® AEROLIZER® consists of a capsule dosage form containing a dry powder formulation of FORADIL (formoterol fumarate) intended for oral inhalation only with the AEROLIZER Inhaler. Each clear, hard gelatin capsule contains a dry powder blend of 12 mcg of formoterol fumarate and 25 mg of lactose (which contains trace levels of milk proteins) as a carrier. Ten capsules are contained in each package, which is clearly labeled. To use the delivery system, a FORADIL capsule is placed in the well of the AEROLIZER Inhaler, and the capsule is pierced by pressing and releasing the buttons on the side of the device. The formoterol fumarate formulation is dispersed into the air stream when the patient inhales rapidly and deeply through the mouthpiece.
  Arms: corticosteroid + long acting beta agonist; steroids
Drug: foradil placebo — open-labeled inhaled corticosteroids (ICS); foradil placebo
  Arms: placebo + corticosteroid + long acting beta agonist; steroids
Drug: foradil — open-labeled inhaled corticosteroids (ICS); foradil
  Arms: corticosteroid + long acting beta agonist; steroids

SUMMARY:
Asthma is the most common chronic disease of childhood affecting 6.2 million children between 2 and 18 years of age, and is the most common cause of school absenteeism due to chronic disease. African American children are 3 to 4 times more likely to be hospitalized for asthma and 4 to 6 times more likely to die from the disease compared to European Americans. The economic burden in this country from asthma is enormous, exceeding $16 billion in 2004. Though there is no cure for asthma, several drugs are available that have been shown to be generally safe and effective in controlling symptoms. Beta 2 agonists are the most commonly used asthma drugs. When inhaled these drugs relax cells in the lungs, which helps patients with asthma breath easier. Two types of beta agonists in use are short-acting beta agonists (SABA) and long-acting beta agonists (LABA). SABA, like albuterol, are used to provide quick relief of chest tightening which help patients to breathe easier. Long-acting beta agonists (LABA) also help patients breathe easier and for a longer period of time. Continued SABA use (for example, inhale albuterol 3 or 4 times a day) is not recommended, and continued LABA use is recommended only if used together with inhaled corticosteroids (ICS). ICS are the most commonly used drug used in asthma that protects against inflammation in the lung. Studies over the past 50 years suggest that continued use of SABA, LABA, and the combination of ICS+LABA may worsen asthma in some patients by reducing the effect of the beta agonists, increasing the rate of asthma attacks, decreasing the ability of the lung to work efficiently, and death. Recent studies suggest asthma worsening by continued beta agonist use occurs in individuals with a certain genotype. Genotype refers to form of the protein, called the beta2 adrenergic receptor (b2AR), in the lung that beta agonists work on. Because of differences in genetic make up, there are different forms of the b2AR. One form is called the Arg16 genotype the other form is called the Gly16 genotype. Compared to Gly16 genotypes, patients with asthma genotyped as Arg16 appear to be more susceptible to asthma worsening that has been associated with continued use SABA, LABA or ICS+LABA. Most of the studies of the influence of genotype on asthma worsening associated with beta agonist use have been performed in adults. The results of a small number of studies suggest children are more susceptible to asthma worsening from chronic beta agonist use compared to adults, and that children with the Arg16 genotype are more susceptible to having asthma attacks than children with the Gly16 genotype. Some evidence suggest that children with asthma should not be treated with ICS+LABA, yet since 2000, the rate at which children with asthma are switched from ICS therapy alone to ICS+LABA has increased significantly. The major question posed by the proposed study is: Does treatment with ICS+LABA compared to ICS alone cause worsening of asthma in children with asthma genotyped as Arg16 homozygotes but not in Gly16 homozygotes? The specific aim of the project is to evaluate the safety of ICS+LABA in children with asthma when separated according genotype. Children with asthma will be screened, be assented and their care taker (parent, for example) consented. A sample of saliva will be collected from which genetic material (DNA) will be collected for the purpose of genotyping. A total of 90 European and African American children, 45 Arg16 and 45 Gly16 genotypes, will be treated for 16 weeks. Half of each genotype will be randomly assigned to receive ICS alone for 16 weeks the other half will receive ICS+LABA. At the end of 16 weeks, those starting with ICS will be then receive ICS+LABA while those who received ICS+LABA first will then take ICS alone. Before and once a month during treatment, each participant will visit the clinic to undergo tests that will assess lung function, how well asthma is being controlled, level of inflammation and quality of life. The results of our study are expected to have a major impact on the way children with asthma are being treated with drugs. If the results of our study show that Arg16 genotypes have worse asthma when they are taking ICS+LABA compared to ICS alone we will conclude that the safety of combination in children is questionable and should be tested in a larger population of children to determine if this popular combination should be used in children with asthma. If the results show that the combination in both genotypes does not worsen asthma compared to ICS treatment, we will conclude that the combination is safe to use in children, at least for 16 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Age of participants will be 5 to 18 yo. FORADIL® is FDA-approved for children in this age group.
* Ethnicity; European and African American will be selected for study. Other minorities will not be studied owing to the problem of population stratification, which refers to differences in allele frequency between cases and controls that are due to differences in ancestry rather than associations of genes with disease or drug response (47). For European Americans, the frequency of Arg16 homozygosity is about 15% compared to about 30% in African Americans (48). In previous studies, the PI restricted his analyses to European Americans because of the potential confounding of population stratification (48;49). .
* Participants must have a diagnosis of asthma. In addition, participants must have persistent asthma as defined by NAEPP guidelines: asthma symptoms > 2 days; > 3 to 4 nighttime awakenings; SABA use >2 days/week; pre-bronchodilator % predicted >60%; FEV1/FVC normal or reduced by 5%.
* Bronchodilator reversibility 12% from baseline; or a history of 12% reversibility during past 12 months; methacholine PC20 < 16 mg/ml.

Exclusion Criteria:

* FEV1< 50% of predicted. Methacholine bronchoprovocation limited to participants with FEV1> 70% of predicted.

  * Other major chronic illnesses: non-skin cancer, cystic fibrosis, bronchiectasis, myelomeningocele, sickle cell anemia, endocrine disease, congenital heart disease, congestive heart failure, stroke, severe hypertension, insulin-dependent diabetes mellitus, renal failure, liver disorders, immunodeficiency state, significant neuro-developmental delay or behavioral disorders (excluding mild attention deficit hyperactivity disorder), or other conditions that would interfere with participation in the study.
  * Participants will discontinue all asthma medications for the duration of the study including theophylline, LTRAs (montelukast), LABA monotherapy, ipratropium bromide. The design of the study ensures that participants will be on ICS (or ICS+LABA) throughout the study and access to SABA for relief.
  * Allergy to methacholine
  * Non-adherence during run-in, or inability or unwillingness of the legal guardian to provide consent or inability or unwillingness of child to provide assent
  * Inability of perform baseline measurements
  * < 80% completion of screening period diaries
  * Inability to contract by telephone
  * Intention to move out of area with 12 months
  * Participants of appropriate age who might be pregnant at time of enrollment will be screened and cannot participant if pregnant.

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2010-10; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Asthma Control Scores will be compared between treatments and genotypes | 16 weeks